CLINICAL TRIAL: NCT03972618
Title: Evaluation of the Efficacy of Sawyer Point One Filters in Schools and Homes in the Dominican Republic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dordt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: DR001
Record Dates: First submitted 2019-05-31; First posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Diarrhea
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- School and village (Experimental): Simultaneous installation of filters in schools and the village
  Interventions: Behavioral: Installation of water filtration system for filtering existing water source
- School only (Experimental): Initial installation in school only
  Interventions: Behavioral: Installation of water filtration system for filtering existing water source
- Village only (Experimental): Initial installation in village only
  Interventions: Behavioral: Installation of water filtration system for filtering existing water source
- Control (No Intervention): Control group. No filter installation initially.

INTERVENTIONS:
Behavioral: Installation of water filtration system for filtering existing water source — Installation of water filtration system and education on hand washing.
  Arms: School and village; School only; Village only

SUMMARY:
Nathan Tintle, in conjunction with others at Dordt College including Dr. Kristin Van De Griend and undergraduate student research assistants, have agreed to collaborate with Hope College to analyze the impact of different water filter deployment strategies in schools and villages on diarrhea and other medical and economic outcomes. The distribution of the water filters will begin in September 2018 to Child Hope schools in 4 different countries (Dominican Republic, Guatemala, Honduras, and Nicaragua). In order to evaluate efficacy of alternative filter deployment strategies, filters will be distributed in 4 separate treatment arms including schools, homes, simultaneous home/school and a control group

DETAILED DESCRIPTION:
Nathan Tintle, in conjunction with others at Dordt College including Dr. Kristin Van De Griend and undergraduate student research assistants, have agreed to collaborate with Hope College and Sawyer Products, Inc. to analyze the impact of different water filter deployment strategies in schools and villages on diarrhea and other medical and economic outcomes. The distribution of the water filters will begin in September 2018 to Child Hope schools in 4 different countries (Dominican Republic, Guatemala, Honduras, and Nicaragua). In order to evaluate efficacy of alternative filter deployment strategies, filters will be distributed in 4 separate treatment arms:

Arm 1: Simultaneous installation of filters in schools and the villages sending children to the school Arm 2: Initial installation of the water filters in a school, with later installation in the corresponding village Arm 3: Instillation of the water filters in villages, with later installation in the corresponding school Arm 4: Control arm. No filter installation initially but, ultimately, installation of filters in both the schools and villages.

Self-reported information on filter usage and health outcomes will be collected through surveys administered to parents (in the households in the villages), teachers (in the schools) and school administrators. Data collection will occur at baseline (when filters are installed), at 2 and 8 weeks post installation. The major goal of this project is to better understand the different health impacts of each different deployment strategy on child and family wellbeing. Better understanding of these filter installation strategies will help guide us as we make filter deployment decisions to provide access to clean drinking water.

ELIGIBILITY:
Inclusion Criteria:

* Lives in selected villages and has children that attend the local school

Exclusion Criteria:

* No children attending the local school

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 698 (Actual)
Dates: Start 2018-09-22 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Diarrhea | 2-weeks
  self-report of diarrhea

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Tintle, Ph.D., Principal Investigator — Dordt College
Locations (1):
- Child Hope Network, Santo Domingo, Dominican Republic

IPD SHARING:
Plan to Share IPD: Undecided
Available upon reasonable request

REFERENCES:
- [Derived] Tintle N, Van De Griend K, Ulrich R, Wade RD, Baar TM, Boven E, Cooper CEA, Couch O, Eekhoff L, Fry B, Goszkowicz GK, Hecksel MA, Heynen A, Laughlin JA, Les SM, Lombard TR, Munson BD, Peterson JM, Schumann E, Settecerri DJ, Spry JE, Summerfield MJ, Sunder M, Wade DR, Zonnefeld CG, Brokus SA, Moen FS, Slater AD, Peterson JW, Pikaart MJ, Krueger BP, Best AA. Diarrhea prevalence in a randomized, controlled prospective trial of point-of-use water filters in homes and schools in the Dominican Republic. Trop Med Health. 2021 Jan 4;49(1):1. doi: 10.1186/s41182-020-00291-y. PMID 33397511